CLINICAL TRIAL: NCT06178601
Title: An Open-label, Single-arm, Multi-center, Phase II Study to Evaluate the Efficacy and Safety of RC48-ADC Combined With AK104 in HER2-expression Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Study of RC48-ADC Combined With Cadonilimab（AK104）in the Treatment of HER2-expression Locally Advanced or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Province Cancer Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-RC48 UC 01
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC plus cadonilimab（AK104） (Experimental): RC48-ADC plus cadonilimab（AK104）
  Interventions: Drug: RC48-ADC; Drug: AK104

INTERVENTIONS:
Drug: RC48-ADC — RC48-ADC （2.0 mg/kg，intravenous (IV) infusion，Q2W）, combined with cadonilimab（AK104）
Drug: AK104 — AK104（6.0 mg/kg，intravenous (IV) infusion，Q2W）combined with RC48-ADC

SUMMARY:
This study will evaluate the efficacy and safety of RC48-ADC combined with AK104 in HER2-expression locally advanced or metastatic urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 6 month.
* Histologically and/or cytologically confirmed locally advanced or metastatic urothelial carcinoma (including urothelial carcinoma originating in the renal pelvis, ureter, bladder, or urethra).
* Pior not received systemic therapy, and can not tolerant cisplatin or refuse chemotherapy.
* HER2 expressing (i.e. IHC 1+ 2+ or 3+) as confirmed by the local lab.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Have at least one evaluable lesion (RECIST 1.1 criteria)
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Has received other antitumor therapy before planned start of trial treatment.
* Previously received allogeneic stem cell or parenchymal organ transplantation;
* Previously or currently suffering from congenital or acquired immunodeficiency diseases;
* known or suspected to have a history of allergies to similar drugs such as RC48-ADC and anti-PD-1, or has a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or is allergic to excipients of the study drug.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* NYHA Class III or IV heart failure.
* Suffering from active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Required systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to enter the trial.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by Investigator | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.

SECONDARY OUTCOMES:
DCR | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
PFS | Up to approximately 30 months
  Progression-free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first.
OS | Up to approximately 40 months
  OS is the time from randomization to death due to any cause safety

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi